CLINICAL TRIAL: NCT05992142
Title: ChAracterizing the Remission Status in Patients With Ulcerative Colitis Treated by 5-ASA
Acronym: CARUC-ASA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIRD2022001; 2022-001683-10 (EudraCT Number)
Record Dates: First submitted 2022-12-13; First posted 2023-08-15 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Ulcerative Colitis
Keywords: remission; 5-aminosalicylate acid (5-ASA)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: transversal study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UC patients (Other): UC patients, treated by 5-ASA for at least 6 months, free of concomitant UC medications for at least 3 months and presenting for a routine follow-up visit
  Interventions: Drug: 5-ASA

INTERVENTIONS:
Drug: 5-ASA — Assessment of the different levels of remission (clinical, endoscopic, histological) in UC patients treated only by 5-ASA, who report to be in clinical remission during a routine follow-up visit

SUMMARY:
For the last years the aim of the management of ulcerative colitis (UC) has become more ambitious including not only clinical remission but also the achievement of biological remission, endoscopic and histological healing, which are associated with less flares, hospitalizations and surgeries. About 50% of the patients with UC followed in routine are treated by 5-aminosalicylate acid (5-ASA) (oral and/or topical). The aim of the study is to describe the different levels of remission (clinical, endoscopic, histological) in UC patients treated only by 5-ASA, that report to be in clinical remission during a routine follow-up visit. The factors associated with different levels of remission (demographic, 5-ASA regimen, biologic, endoscopic, histologic) will be studied. Adherence and quality of life will be examined through patient questionnaires.

DETAILED DESCRIPTION:
The management of inflammatory bowel diseases aims to induce not only a clinical corticosteroid-free remission but also a deep remission defined by the achievement of mucosal healing. In ulcerative colitis (UC), mucosal healing has been nicely correlated with a better outcome of the disease. A lack of mucosal healing after a first steroid course is associated with a bad outcome including higher hospitalizations and more clinical relapses after 1 year. The absence of mucosal healing has also been correlated with higher rates of colectomy. Mucosal healing is defined by the absence of ulcers and includes patients with an endoscopic Mayo subscore of zero and one. Recently, a significantly better outcome has been demonstrated in patients having an endoscopic Mayo subscore of zero instead of one as well as a histological healing on the biopsies. The fecal biomarkers, especially the fecal calprotectin, have a high accuracy for the prediction of ongoing endoscopic and histologic inflammation in patients in clinical remission. Fecal calprotectin is well correlated with the Mayo endoscopic subscore and can discriminate patients with an endoscopic Mayo subscore of zero versus one or more by using a cut-off of 150 microgram/gram. A residual histologic inflammation is associated with a fecal calprotectin of 155 microgram/gram or more. Subsequently the management of UC has evolved and aims to induce a tighter control of the disease including a complete endoscopic response and a histological healing. It is currently not known how well these patients who report being in clinical remission are actually in objectively defined remission. As a deep remission is so important for the future evaluation of the disease, it is important to understand the factors linked to the absence of such remission.

The primary objective of this study is to describe the percentage of the different levels of remission (clinical, endoscopic, histological), in UC patients, treated by 5-ASA for at least 6 months, free of concomitant UC medications for at least 3 months and presenting for a routine follow-up visit.

The secondary objectives of this study are:

* to identify the factors associated to the absence of deep remission (demographic, UC history, clinical, biological, endoscopic, histological, 5-ASA regimen, adherence)
* to describe the adherence of the patients to the 5-ASA medications and its impact on the remission status.
* to describe the regimen of 5-ASA prescription (dosage, oral/local form) and its impact on the remission status.
* to describe the quality of life of the patients with UC on 5-ASA and its correlation with the level of remission.
* to understand the implication of patient's perspective and physician's perspective in patient lacking deep remission.
* to analyze the reasons of non-deep remission

This study is a national, multicenter, transversal, interventional study conducted in Belgium (16 centers will participate). The trial design is as follows:

* All subjects will undergo screening procedures. The screening visit of eligible patients will include the review of inclusion and exclusion criteria, and the informed consent form procedure. After screening, if the patient fulfils all inclusion and none of the exclusion criteria, and is willing to participate, the inclusion visit will be performed at the same time. The gastroenterologist will record the characteristics of patients and of the disease, medical history, current and past UC treatments in the last year before inclusion, and the PRO-2 score and bowel urgency in the last 3 days before the visit.
* A sigmoidoscopy with 2 biopsies (taken in the most inflamed area) as well as a fecal calprotectin measurement will be performed during the inclusion visit. The sigmoidoscopy procedure will be scored locally by the gastroenterologist with the endoscopic Mayo score and the UCEIS score. The Geboes score will be calculated centrally.
* The patient will complete the Short Health Scale and the Medication Adherence Report Scale.
* Biochemistry (including hematocrit, hemoglobin, platelets count, leucocytes, CRP, urea and serum creatinine) is not obligatory, but if it is planned in the routine management of the patient, these data will be recorded for study purposes.
* In patients not achieving complete endoscopic remission (Endoscopic Mayo subscore >0), an exploratory questionnaire will be answered by the physician about "physician perspective" regarding the treatment strategy to explore the supposed reasons of the absence of UC remission. Depending on the answer, an exploratory questionnaire can be directed towards the patient exploring the reason for possible low adherence or deliberately refusing other medications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Confirmed diagnosis of UC
3. Patients with PRO-2 ≤ 1, with ≤ 1 for stool frequency and 0 for rectal bleeding in the last 3 days before the visit.
4. Recruitment during a routine follow-up visit.
5. Subjects to whom 5-ASA treatment has been prescribed for at least 6 months (any type of oral and/or rectal 5 ASA, any dosage) and with the dose of 5-ASA stable for at least 2 weeks (including suppositories) prior to inclusion.
6. Prescription of 5-ASA is within the locally approved Summary of Product Characteristics (SmPCs)
7. Subjects free of concomitant UC medication (corticosteroids, immunomodulators, biologics, JAK inhibitors, S1PR modulator or investigational drugs) for at least 3 months
8. Subject or the subject's legally acceptable representative have the capacity to understand and (voluntary) sign an informed consent form
9. Be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

Any subject who meets one of the following criteria will not qualify for entry in the study:

1. Subjects currently treated by immunomodulators, biologics, JAK inhibitors, S1PR modulator and investigational drugs and within the last three months. A history of immunomodulator or biologic or JAK inhibitor or S1PR modulator and investigational drugs use in the past is not an exclusion criteria.
2. Subjects recruited during hospitalization, or via the urgency department for active UC, or during an unscheduled visit for emergency reasons.
3. UC patients with a total colectomy, with or without IPAA
4. Patients with indetermined colitis (IBDU)
5. Women that are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Complete clinical remission | week 0
  Complete clinical remission is defined by a PRO-2 = 0 and no bowel urgency
Endoscopic remission | week 0
  Endoscopic remission is defined by an endoscopic MAYO subscore of 0 or 1 and/or by a Ulcerative Colitis Endoscopic Index of Severity (UCEIS) of 0 or 1
Histological remission | week 0
  Histological remission will be defined by the absence of any acute inflammatory activity on the biopsies according to the Geboes score, including Geboes 0-1
Deep remission | week 0
  Deep remission will be defined by the combination of complete clinical, complete endoscopic and histological remission

SECONDARY OUTCOMES:
Demographic factors associated to the absence of deep remission | week 0
  Demographic factors questionnaire: year of birth, sex (male/female), ethnic origin (Caucasian/Black/Hispanic/Asian/Other) and smoking status (Smoker with > 1 cigarette/day, Non-smoker or Former smoker)
Disease characteristics associated to the absence of deep remission | week 0
  Disease characteristics questionnaire: diagnosis date ('DD-MMMM-YYYY') and UC Montreal classification [E1 (Ulcerative proctitis), E2 (left-sided UC), E3 (Extensive) or Pancolitis]
Medical history associated to the absence of deep remission | week 0
  Medical history questionnaire with a list of current and past concomitant medical conditions including extra-intestinal manifestations (yes/no)
Medication history associated to the absence of deep remission | week 0
  A questionnaire (yes/no) about UC medication history prescribed the year before inclusion and current medication use including corticosteroids including local forms, immunomodulators, biologics, JAK inhibitors, S1PR modulator or investigational drugs): brand name, date of start and stop, frequency, route of administration and dosage. Details on past and current 5-ASA use will be recorded: brand name, date of start and stop, formulation (oral, rectal, enema), dosage, frequency.
Disease activity based on PRO-2 score associated to the absence of deep remission | week 0
  Disease activity measurement based on Two component Patient Reported Outcome (PRO-2) score (stool frequency and rectal bleeding; average score of the last 3 days before the visit), using a grading scale from 0 (normal) to 3 (for rectal bleeding: blood alone passed and for stool frequency: >= 5 stools more than normal)
Disease activity based on bowel urgency associated to the absence of deep remission | week 0
  Disease activity measurement based on bowel urgency for the past 24 hours using a VAS scale from 0 (no urgency) to 10 (worst possible urgency)
Disease activity based on endoscopic score associated to the absence of deep remission | week 0
  Disease activity measurement based on Mayo and UCEIS endoscopic score, using a grading scale from 0 (normal/inactive) to 3 (active)
Disease activity based on histological Geboes score associated to the absence of deep remission | week 0
  Disease activity measurements based on histological Geboes score, with grade 0-1=inactive/absent, grade 2= chronic inflammation and grade 3-5 = acute inflammation
Disease activity based on objective markers associated to the absence of deep remission | week 0
  Disease activity measurement based on the objective markers fecal calprotectine value (microg/g) and C-reactive protein (CRP) value (mg/L) if available
Adherence associated to the absence of deep remission | week 0
  Adherence based on Medication Adherence Report Scale (MARS-5)
The percentage of adherent patients on 5-ASA medications | week 0
  The percentage of adherent patients on 5-ASA medications, and an adherent patient is defined by a total Medication Adherence Report Scale (MARS-5) score of 21 or by a MARS-5 score of 4 for each individual question.
The impact of adherence on the remission status | week 0
  The percentage of adherent patients on 5-ASA medications will be compared between the different levels of remission (clinical remission, endoscopic remission, histological remission, deep remission, non-deep remission)
The percentage of prescription of the different 5-ASA regimens | week 0
  The percentage of prescription of the different 5-ASA regimens, and the prescription rate of the different 5-ASA regimens depends on the dosage (grams), oral and/or topical form.
The impact of the prescription rate of the different 5-ASA regimens on the remission status | week 0
  The prescription rate of the different 5-ASA regimens will be compared between the different levels of remission (clinical remission, endoscopic remission, histological remission, deep remission, non-deep remission)
Quantification of the quality of life of the patients with UC on 5-ASA | week 0
  Quality of life based on validated Short Health Scale (a four-part visual analogue scale questionnaire using open-ended questions that are designed to assess the impact of IBD on a health related quality of life, with score between 0 and 40; lower score, better quality of life)).
Correlation of the quality of life scores with the level of remission | week 0
  Quality of life scores will be correlated with the different levels of remission (clinical remission, endoscopic remission, histological remission, deep remission, non-deep remission)
The factors associated with non-deep remission coming from either physician management or patient perception | week 0
  In patients not achieving complete endoscopic remission (Endoscopic Mayo subscore >0), an exploratory questionnaire will be answered by the physician about "physician perspective" regarding the treatment strategy to explore the supposed reasons of the absence of UC remission. Depending on the answer, an exploratory questionnaire can be directed towards the patient exploring the reason for possible low adherence or deliberately refusing other medications.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Reenaers, MD, PhD, Principal Investigator — Study Principal Investigator
Locations (16):
- Belgium (16):
  - Imelda Ziekenhuis, Bonheiden
  - Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Sint-Lucas Gent, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHU de Liège - Site Sart Tilman, Liège
  - Groupe santé CHC Clinique du MontLégia, Liège
  - AZ Voorkempen Malle, Malle
  - AZ Damiaan, Ostend
  - AZ Delta, Roeselare
  - Sint-Andries ziekenhuis Tielt, Tielt
  - AZ Vesalius, Tongeren
  - AZ Turnhout, Turnhout
  - CHU UCL Namur -Site Mont Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BIRD website — https://www.birdgroup.be/en